CLINICAL TRIAL: NCT02957708
Title: Effectiveness of Modified Constraint-induced Movement Therapy and Self-regulation Learning for Children With Hemiplegic Cerebral Palsy
Brief Title: Constraint-induced Movement Therapy and Self-regulation for Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Western Sydney (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Karen Liu, Associate Professor, University of Western Sydney
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SR-CIMT_CP
Record Dates: First submitted 2016-09-22; First posted 2016-11-08 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mCIMT + SR (Experimental): modified constraint-induced movement therapy plus self regulation
  Interventions: Other: mCIMT + SR
- Control (Active Comparator): conventional occupational therapy
  Interventions: Other: Control

INTERVENTIONS:
Other: mCIMT + SR — Each participant wears a customized cotton sling on the unaffected arm for six hours everyday. Participant is engaged in fifteen unimanual tasks during the three-week training that provides them sufficient challenge and opportunities for repetition.
  SR is incorporated on the 1-hour structured practice by using video playback to help participants realize their own performance for better learning. Participant first performs a task with videotaping, then identifies steps with problems or difficulties by video playback of participant's performance. Secondly, participant is asked for possible solutions, prompting is given if needed. Lastly, participant performs the activity by adopting the suggested solutions with videotaping again to facilitate participant's evaluation of new performance.
  Arms: mCIMT + SR
Other: Control — A combination of training on functional and remedial activities on unimanual tasks and bimanual tasks that based primarily on neurodevelopmental approach are provided. The training aims at increasing control, strength and functional use of their affected arm and hand, and improving bimanual coordination in performing daily activities. Each participant receives 1 to 2 hours of training per week at school. Home exercise including both unimanual and bimanual tasks is prescribed to them as well.
  Other Names: Conventional occupational therapy
  Arms: Control

SUMMARY:
This study examines the effect of combining modified constraint-induced movement therapy (mCIMT) and self-regulation (SR) in promoting upper limb function of children with hemiplegic cerebral palsy (CP) studying in a school-based setting.

DETAILED DESCRIPTION:
Children diagnosed with hemiplegic CP are involved. A within-subject design is used with children acting as their own controls. The study is scheduled at three-week intervals. All children undergo conventional occupational therapy (OT) and modified constraint-induced movement therapy plus self-regulation (mCIMT + SR) program in a random order.

Both programs last for three weeks. Each program is followed by a three-week no-treatment period to measure the carry-over effect. The OT program consists of training on unimanual and bimanual tasks for 1 to 2 hours a week with daily home exercise. The mCIMT + SR program involves restraint of the unaffected upper limb of children using a cotton sling for 6 hours per day for 15 days. A one-hour structured task practice with the use of SR is provided during each 6-hour restraint.

The Bruininks-Oseretsky Test of Motor Proficiency, the Jebsen-Taylor Test of Hand Function, the Caregiver Functional Use Survey, a hand dynamometer, pinch gauge, and modified Ashworth scale are used for evaluation. All children are assessed for five times at 3-week interval: once before and twice after the conventional OT; and twice after the mCIMT + SR at 1 week and at 3 weeks.

Before and after the three-week intervention, the children participate in event-related potentials (ERP) sessions with a choice reaction task. Event-related potentials (ERP) technique is used to capture the changes in neural mechanism after intervention.

ELIGIBILITY:
Inclusion Criteria:

* children with diagnosis of hemiplegic CP,
* 6-18 years of age studying at local special school for students with physical handicap (PH),
* intelligence ranging from normal to mild grade mental retardation,
* the ability to extend the wrist at least 20° and the metacarpophalangeal joint 10° from full flexion, and
* no balance problems sufficient to compromise safety.

Exclusion Criteria:

* any health problems that were not associated with CP, and
* severe muscle tone with modified Ashworth scale scored greater than 3.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2007-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Change in Bruininks-Oseretsky Test of Motor Proficiency | Assessment 1 (before intervention 1); Assessment 2 (after intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (after intervention 2); Assessment 5 (3 weeks after no treatment) (refer to description)
  Subtest 5 ((upper-limb coordination) and subtext 8 (speed and dexterity), testing the upper limb function are used.
  Time frame:
  Assessment 1 (within two days before intervention 1); Assessment 2 (within two days after the three-week intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (two days after the three-week intervention 2); Assessment 5 (3 weeks after no treatment)
Change in Jebsen-Taylor Test of Hand Funcion | Assessment 1 (before intervention 1); Assessment 2 (after intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (after intervention 2); Assessment 5 (3 weeks after no treatment) (refer to description)
  It assesses hand function using seven unimanual tasks: writing, turning cards over, picking up small commonly encountered objects, simulated eating, stacking checker, and moving light and heavy cans.
  Time frame:
  Assessment 1 (within two days before intervention 1); Assessment 2 (within two days after the three-week intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (two days after the three-week intervention 2); Assessment 5 (3 weeks after no treatment)

SECONDARY OUTCOMES:
Change in Caregiver Functional Use Survey | Assessment 1 (before intervention 1); Assessment 2 (after intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (after intervention 2); Assessment 5 (3 weeks after no treatment) (refer to description)
  It reviews caregivers' perceptions of how much and how well their child use the affected upper limb in the real-life situation.
  Time frame:
  Assessment 1 (within two days before intervention 1); Assessment 2 (within two days after the three-week intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (two days after the three-week intervention 2); Assessment 5 (3 weeks after no treatment)
Change in Grip strength | Assessment 1 (before intervention 1); Assessment 2 (after intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (after intervention 2); Assessment 5 (3 weeks after no treatment) (refer to description)
  It is measured using a Jamar hand dynamometer.
  Time frame:
  Assessment 1 (within two days before intervention 1); Assessment 2 (within two days after the three-week intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (two days after the three-week intervention 2); Assessment 5 (3 weeks after no treatment)
Change in Pinch strength | Assessment 1 (before intervention 1); Assessment 2 (after intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (after intervention 2); Assessment 5 (3 weeks after no treatment) (refer to description)
  It is measured using a pinch gauge.
  Time frame:
  Assessment 1 (within two days before intervention 1); Assessment 2 (within two days after the three-week intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (two days after the three-week intervention 2); Assessment 5 (3 weeks after no treatment)
Change in Modified Ashworth scale | Assessment 1 (before intervention 1); Assessment 2 (after intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (after intervention 2); Assessment 5 (3 weeks after no treatment) (refer to description)
  It assesses muscle tone at the shoulder, elbow and wrist.
  Time frame:
  Assessment 1 (within two days before intervention 1); Assessment 2 (within two days after the three-week intervention 1); Assessment 3 (3 weeks after no treatment period and before intervention 2); Assessment 4 (two days after the three-week intervention 2); Assessment 5 (3 weeks after no treatment)

OTHER OUTCOMES:
Change in Choice reaction task | Two days before and two days after the three-week mCIMT + SR intervention
  The children respond by pressing the buttons on an oversized number pad with keys specifying for pressing with the index finger or the thumb. Stimuli are pictures of an outlined hand with responding digit highlighted. When the child sees a thumb highlighted, he or she is required to press the thumb key with the thumb. Alternatively, he or she will press the index finger key with the index finger if the index finger is highlighted in the picture.
  Event-related potentials (ERPs) are recorded from a 64-channel array of electrodes placed in an extended 10-20 system.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hong Kong Polytechnic University, Hong Kong, Hong Kong